CLINICAL TRIAL: NCT02011802
Title: Sorbact TM: Effect of a Microbial Binding Dressing on Wound Healing After Pilonidal Sinus Excision
Acronym: SORKYSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: INRESA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5568
Record Dates: First submitted 2013-10-10; First posted 2013-12-13 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sinus Pilonidal
Keywords: Sorbact TM; Alginates; Dressing; Wound healing
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algosteril TM (Active Comparator): Calcium alginate dressings are made from seaweed. Calcium alginate dressings form a natural gel of the exudates against the healing tissue that keeps it moist and supple, aiding in healing and tissue growth. In addition, this gel material forms a natural barrier to bacteria that may complicate healing with secondary infections of the wound. Alginates are the reference of dressing after sinus pilonidal excision.
  Interventions: Device: Algosteril TM
- Sorbact TM (Experimental): DACC (dialkylcarbamoyle chloride) is a main component of the bacterial binding wound dressing: Sorbact. DACC is a hydrophobic fatty acid derivative that can be used to coat dressing materials, resulting in a dressing with highly hydrophobic pathogen binding properties. This is a primary wound interface dressing and is effective when in close contact with the wound bed in a moist environment.
  Interventions: Device: Sorbact TM

INTERVENTIONS:
Device: Algosteril TM
  Arms: Algosteril TM
Device: Sorbact TM
  Arms: Sorbact TM

SUMMARY:
Sinus pilonidal concern 26/100 000 young adults. It manifests after puberty, presenting as an acute abscess in approximately 50% of patients or as a discharging painful sinus. Patients may experience lengthy healing times resulting in considerable morbidity and disruption to a young adult's life. Eradication of pilonidal sinus is based on a wide surgical excision and at the end of the procedure, the wound is dressed with an alginate dressing (Algosteril®).

The objective is to show a better efficiency of Sorbact TM (trademark) dressings compared to Alginates that are standardized dressings after pilonidal sinus excision during a period of 75 days. The main objective is to show a difference of 20% of wounds completely healed in 75 days between the two types of dressing: 50% of wounds healed with Algosteril TM compared to 70% of wounds healed with Sorbact TM.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old
* Informed consent signed by the participant
* Affiliation to social security system
* Having a pilonidal sinus:

  * Asymptomatic or discovered by the patient during a routine examination
  * With chronic recurrent infection and skin rupture

Exclusion Criteria:

* Patients with concomitant pathology:

  * cancer treated by chemotherapy
  * Hypertension uncontrolled systolic blood pressure>180 mmHg or diastolic> 110 mmHg
  * Severe comorbidity with reduced life expectancy less than 12 months
  * Acute cardiovascular disease (myocardial infarction, stroke, recent heart surgery) within 3 months before inclusion
* Patients participating in another clinical trial
* Known for intolerance to one of the dressings
* Known pregnancy
* Uncontrolled diabetes (fasting glucose >2g/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of wounds healed | 75 days after surgery

SECONDARY OUTCOMES:
Total surface area measure of non-healed wounds | 75 days after surgery
VAS pain | every 2 weeks, from randomization up to 4 months or date of healing, whichever comes first
analgesic use | every 2 weeks, from randomization up to 4 months or date of healing, whichever comes first
antibiotics use | every 2 weeks, from randomization up to 4 months or date of healing, whichever comes first
number of dressings used | every 2 weeks, from randomization up to 4 months or date of healing, whichever comes first

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de Chirurgie Digestive-Hôpital Pasteur-39 av de la Liberté, Colmar
  - Service de Chirurgie Digestive-Centre Hospitalier de Mulhouse- 20 av du Dr René Laennec, Mulhouse
  - Service de Chirurgie Générale Viscérale et Digestive-Centre Hospitalier de Saverne-19 Côte de Saverne, Saverne
  - Service de Chirurgie Digestive - Hôpital de Hautepierre- Hôpitaux Universitaires de Strasbourg - France, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Romain B, Mielcarek M, Delhorme JB, Meyer N, Brigand C, Rohr S; SORKYSA group. Dialkylcarbamoyl chloride-coated versus alginate dressings after pilonidal sinus excision: a randomized clinical trial (SORKYSA study). BJS Open. 2020 Apr;4(2):225-231. doi: 10.1002/bjs5.50259. Epub 2020 Feb 4. PMID 32020765